CLINICAL TRIAL: NCT06161090
Title: Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of CM310 Recombinant Humanized Monoclonal Antibody Injection in Healthy Subjects
Brief Title: Study of CM310 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310HV001
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 75 mg (Experimental): CM310 Recombinant Humanized Monoclonal Antibody Injection
  Interventions: Biological: CM310
- Group 150 mg (Experimental): CM310 Recombinant Humanized Monoclonal Antibody Injection
  Interventions: Biological: CM310
- Group 300 mg (Experimental): CM310 Recombinant Humanized Monoclonal Antibody Injection
  Interventions: Biological: CM310
- Group 600 mg (Experimental): CM310 Recombinant Humanized Monoclonal Antibody Injection
  Interventions: Biological: CM310
- Placebo (Placebo Comparator): Placebo, Subcutaneous
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CM310 — CM310 injection
  Arms: Group 150 mg; Group 300 mg; Group 600 mg; Group 75 mg
Drug: Placebo — subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a single center, randomized, double-blind, placebo-controlled, dose escalation study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers.
* aged ≥ 18 and ≤ 65 years old.
* With all clinical laboratory examination normal.
* Voluntary signing of the informed consent form.

Exclusion Criteria:

* With a history of asthma and allergic reactions.
* With a history of conjunctivitis and keratitis, as well as previous medical conditions.
* With positive results from alcohol breath or urine drug abuse testing.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Adverse event | up to Week 9
  Incidence of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- PKUCare Luzhong Hospital, Zibo, China

REFERENCES:
- [Derived] Zhang L, Zhang W, Xu Y, Dong L, Sun Y, Jia Y, Li Z, Chen B, Hou J, Zhang J. Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Stapokibart in Healthy Volunteers and Adult Subjects with Atopic Dermatitis. Adv Ther. 2024 Jul;41(7):2953-2965. doi: 10.1007/s12325-024-02887-w. Epub 2024 Jun 4. PMID 38833140